CLINICAL TRIAL: NCT04130477
Title: Computer Designed and Chairside Fabricated Custom Tunnel Attachments Paired With Clear Aligners Versus Traditional Clear Aligners for Orthodontic Leveling and Aligning- A Randomized Controlled Clinical Trial
Brief Title: Tunnel Attachments With Clear Aligners vs Clear Aligners
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harvard School of Dental Medicine (Other)
Responsible Party: Principal Investigator, Alyaa Aldohan, Orthodontic resident and Doctor of Medical Sciences candidate, Harvard School of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HarvardSDM
Record Dates: First submitted 2019-10-10; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: Tunnel attachments as an auxiliary with clear aligners
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Clear aligners with tunnel attachment (Experimental): Participants will receive traditional clear aligner therapy with virtual set up and will be supplemented by virtually planned tunnel attachments which will be threaded by a light Nickel-Titanium wire
  Interventions: Device: Tunnel attachments and light Nickel Titanium wire
- Clear aligners (Active Comparator): Participants will receive traditional clear aligner therapy with virtual set up
  Interventions: Device: Clear Aligner therapy

INTERVENTIONS:
Device: Tunnel attachments and light Nickel Titanium wire — Tunnel attachments planned virtually and light Nickel Titanium wire
  Arms: Clear aligners with tunnel attachment
Device: Clear Aligner therapy — Clear Aligner therapy
  Arms: Clear aligners

SUMMARY:
Incorporating wire threaded custom tunnel attachments with clear aligner therapy is a novel approach developed to address the shortcomings of the currently available orthodontic systems. This hybrid system is anticipated to take advantage of the benefits and overcome many of the limitations of traditional fixed buccal/lingual appliances and clear aligner therapy. The concept utilizes light arch wires to be threaded through computer designed, chairside-fabricated composite tunnel attachments to achieve better control of three-dimensional tooth movements not achievable by clear aligners, such as Invisalign® (Align Technology, Santa Clara, CA) alone. The superelastic feature of the arch wires allows delivery of more continuous forces than aligners alone, potentially permitting shorter duration of recommended aligner wear during orthodontic treatment. A virtual set-up would be used to plan the desired position of the teeth, which in turn will be used to customize the size and position of composite tunnel attachments based on how two round arch wires will pass through tubes within the attachments. The attachments can be placed on either the buccal or lingual surfaces of teeth, depending on clinical preferences and esthetic demands. This is achievable using in-house aligners, which will also allow the fabrication of aligners in the office or at a conventional orthodontic lab at a fraction of the cost of traditional clear aligners.

DETAILED DESCRIPTION:
Specific aims:

* Test and formally describe a novel method that utilizes clear aligners paired with computer-designed, chairside-fabricated tunnel attachments to achieve tooth movements that are challenging for clear aligners.
* Conduct a randomized clinical trial to compare the ability of a traditional clear aligner system Invisalign® (Align Technology, Santa Clara, CA) and a clear aligner system incorporating wire threaded tunnel attachments in:

  * achieving predicted outcomes; discrepancies in bucco-lingual and inciso-gingival positions between the virtual plan and end of treatment intraoral scan and will be measured in millimeters and angular discrepancies will be measured in degrees
  * end of treatment ABO leveling and alignment objective grading scores

Materials and Methods:

A virtual set-up is completed by the clinician to plan the position, orientation, and dimension will be customized on the teeth to be moved.Generally, they are spherically shaped and their dimensions are approximately 2-3 mm. Vacuum-formed attachment template will be made to take the shape of a tube-holding spheres, in which tubes are embedded. The tubes are standard in size with an outside diameter of 0.032", and an inside diameter of 0.019" and 2 mm length The template will be loaded with composite after inserting the metal tubes are placed in their predetermined location on the tray. Double tubes will be used when torque control is needed. 0.016" buccal or lingual round wires will be placed into the tunnel attachments along the attachments. Aligners will be delivered to patient to be worn for at least 8 hours a day and changed as determined by the Dental Monitoring application.

ELIGIBILITY:
Inclusion Criteria:

1. healthy subjects over the age of 10 years and below 65;
2. eruption of all permanent anterior teeth;
3. non-extraction treatment;
4. maximum of 7mm of crowding/spacing;
5. no more than 45 degrees of rotations
6. no more than 7 mm crowding

Exclusion Criteria:

1. presence of systemic diseases, cleft lip and palate, craniofacial anomalies, syndromes affecting bone or teeth, impacted teeth (excluding 3rd molars), congenitally missing lateral incisors, and tumors of the parathyroid gland;
2. the presence of bridges or implants replacing anterior teeth;
3. cases requiring orthognathic surgery;
4. significant (> moderate) periodontal disease, intake of drugs affecting tooth movement or bone formation (chronic use of Non-Steroidal Anti-Inflammatory Drugs, bisphosphonates, levothyroxine, or teriparatide drug class), pregnancy;
5. cases requiring tooth extractions

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
1) Horizontal movement in millimeters | 3-12 months of orthodontic treatment
  The virtual setups (predicted results) and actual results scans will be superimposed using a best-fit alignment method using Geomagic Control X (3D Systems, Rock Hill, South Carolina). Initial alignment will be done using 300 surface points, and fine adjustments will be made using additional 1500 points. This process will be repeated as necessary. Once satisfactory superimposition is performed, the x, y, z coordinates (mm) of dental landmarks on the setup and result arches will be exported and analyzed. Linear and angular measurements will be made to determine the accuracy of each system in achieving predicted vertical, in-out and torque treatment outcomes. The percentage of accurate tooth movement will be determined with the following equation: [(|predicted-achieved|/|predicted|) 100%]
2) Vertical movement in mm | 3-12 months of orthodontic treatment
  The virtual setups (predicted results) and actual results scans will be superimposed using a best-fit alignment method using Geomagic Control X (3D Systems, Rock Hill, South Carolina). Initial alignment will be done using 300 surface points, and fine adjustments will be made using additional 1500 points. This process will be repeated as necessary. Once satisfactory superimposition is performed, the x, y, z coordinates (mm) of dental landmarks on the setup and result arches will be exported and analyzed. Linear and angular measurements will be made to determine the accuracy of each system in achieving predicted vertical, in-out and torque treatment outcomes. The percentage of accurate tooth movement will be determined with the following equation: [(|predicted-achieved|/|predicted|) 100%]
3) angular movement in degrees | 3-12 months of orthodontic treatment
  The virtual setups (predicted results) and actual results scans will be superimposed using a best-fit alignment method using Geomagic Control X (3D Systems, Rock Hill, South Carolina). Initial alignment will be done using 300 surface points, and fine adjustments will be made using additional 1500 points. This process will be repeated as necessary. Once satisfactory superimposition is performed, the x, y, z coordinates (mm) of dental landmarks on the setup and result arches will be exported and analyzed. Linear and angular measurements will be made to determine the accuracy of each system in achieving predicted vertical, in-out and torque treatment outcomes. The percentage of accurate tooth movement will be determined with the following equation: [(|predicted-achieved|/|predicted|) 100%]

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Masoud, BDS, DMSc, Principal Investigator — Harvard School of Dental Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Papadimitriou A, Mousoulea S, Gkantidis N, Kloukos D. Clinical effectiveness of Invisalign(R) orthodontic treatment: a systematic review. Prog Orthod. 2018 Sep 28;19(1):37. doi: 10.1186/s40510-018-0235-z. PMID 30264270
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=Papadimitriou%2C+A.%2C+et+al.%2C+Clinical+effectiveness+of+Invisalign(R)+orthodontic+treatment%3A+a+systematic+review